CLINICAL TRIAL: NCT03085550
Title: A Randomised Controlled Trial to Compare Platelet-Rich Plasma and Autologous Fat Graft for Diabetic Ulcer
Brief Title: Platelet Rich Plasma and Autologous Fat Graft for Diabetic Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/LO/2261
Record Dates: First submitted 2017-03-01; First posted 2017-03-21 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus Foot Ulcer
Keywords: diabetic foot ulcer; diabetes mellitus; fat grafting; platelet rich plasma; wound healing
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Conventional dressings management
- Fat grafting only (Experimental): Patients will undergo conventional fat harvesting as per Coleman technique and infiltration of fat into diabetic ulcer wound bed in 1cc:10cm2 fat:wound size ratio
  Interventions: Procedure: Fat grafting
- Fat grafting + Platelet rich plasma (Experimental): Patients will undergo conventional fat harvesting as per Coleman technique. Fat will be mixed with autologous PRP and infiltrated into diabetic ulcer wound bed in 1cc:10cm2 fat:wound size ratio
  Interventions: Procedure: Fat grafting + platelet rich plasma

INTERVENTIONS:
Procedure: Fat grafting — Single treatment fat grafting infiltrated into diabetic ulcer wound
  Arms: Fat grafting only
Procedure: Fat grafting + platelet rich plasma — Single treatment fat grafting mixed with autologous platelet rich plasma infiltrated into diabetic ulcer wound. Autologous PRP is obtained using the ANGEL(TM) Concentrated Platelet Rich Plasma (cPRP) Separation Device which is FDA-regulated and CE certified
  Arms: Fat grafting + Platelet rich plasma

SUMMARY:
Conventional management of diabetic ulcers is associated with slow healing, high costs and repeated trips to clinic. Stem cells contained in fat grafts can differentiate into pro-healing cells and release growth factors with evidence suggesting a benefit in wound healing. Platelet-rich-plasma (PRP), an autologous blood-product, demonstrates pro-healing properties through releasing pro-healing factors and regulating angiogenesis. When used combination there is evidence of additional wound healing benefits.

The aim is to investigate the feasibility of conducting a randomised controlled trial with fat grafting and fat/PRP co-grafting as interventions for diabetic ulcers. We aim to develop pilot data which can power a multi-centre study. The aim of the trial would be to determine the feasibility of the trial by assessing recruitment, randomisation and retention of participants. We would also evaluate the rate of wound healing in diabetic ulcers when treated with conventional dressings, fat grafting alone and fat+PRP combination. The secondary aims will be to understand the mechanism of the healing process, the health related quality of life and patient satisfaction and the cost implications.

The study is a single-blinded randomised controlled trial of approximately 30 patients with three parallel treatment arms. Each patient will be followed up for 12 weeks and the rate and degree of wound healing will be assessed. Wound biopsies will be taken at Day 0, week 1 and week 4 and will undergo subsequent histological analysis to evaluate the mechanism of healing. The study is expected to last two years from recruitment of the first patient and will be conducted at Royal Free Hospital and UCL Division of Surgery and Interventional Science.

The combination of fat+PRP may provide diabetic patients the option of a single treatment with improved healing, shorter followup and a reduced cost burden. Validation of the mechanism of healing through histological analysis will confirm clinical findings and help guide future research.

DETAILED DESCRIPTION:
RCT to compare fat grafting and fat grafting with PRP in chronic diabetic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 18-90 at the time of consent;
* Diabetic foot ulcer (DFU) measuring more than 0.5cm x 0.5cm and less than 10cm x 10cm;
* Wound with clean, healthy granulating bed, with minimal adherent slough;
* Patient understands and is willing to participate and can comply with weekly visits and follow-up regime.

Exclusion Criteria:

* Wound with active infection;
* Patients with underlying vascular insufficiency (ABPI<0.3);
* Uncontrolled Diabetes Mellitus, as measured by an HbA1c > 90mmol/mol;
* Presence of one or more medical conditions, including renal, hepatic, haematologic, active auto-immune or immune diseases that, would make the subject an inappropriate candidate for this ulcer healing study;
* Patient not fit for surgery (ASA classification > 4).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Rate of wound healing | 12 weeks
  Comparison of rate of wound healing between each group
Degree of wound healing | 12 weeks
  Comparison of degree of wound healing (50% and 100% re-epithelialisation)

SECONDARY OUTCOMES:
Mechanism of wound healing | 12 weeks
  Histological analysis of wound biopsies from each group at day 0, week 1 and week 4
Health related quality of life | 12 weeks
  Patient quality of life with each procedure
Cost implications | 12 weeks
  Cost implications of each treatment arm as per NHS coding practice
Patient reported outcome measures | 12 weeks
  Patient reported outcome measures of satisfaction of each procedure

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Smith, MBChB, Principal Investigator — University College, London
Locations (1):
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Nolan GS, Smith OJ, Heavey S, Jell G, Mosahebi A. Histological analysis of fat grafting with platelet-rich plasma for diabetic foot ulcers-A randomised controlled trial. Int Wound J. 2022 Feb;19(2):389-398. doi: 10.1111/iwj.13640. Epub 2021 Jun 24. PMID 34169656
- [Derived] Smith OJ, Leigh R, Kanapathy M, Macneal P, Jell G, Hachach-Haram N, Mann H, Mosahebi A. Fat grafting and platelet-rich plasma for the treatment of diabetic foot ulcers: A feasibility-randomised controlled trial. Int Wound J. 2020 Dec;17(6):1578-1594. doi: 10.1111/iwj.13433. Epub 2020 Jul 7. PMID 32633854